CLINICAL TRIAL: NCT01404546
Title: A Randomized Controlled Pilot Study of Standardized Counselling and Cost-free Pharmacotherapy for Smoking Cessation Among Stroke and TIA Patients
Brief Title: Cost Free Pharmacotherapy for Smoking Cessation in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Sophia Papadakis, Associate Professor, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UOHI2010-1
Record Dates: First submitted 2011-07-26; First posted 2011-07-28 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2011-07

CONDITIONS: Stroke
Keywords: stroke smoking cessation cost-free pharmacotherapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cost Free Pharmacotherapy (Experimental): Participants assigned to the CF group received a starter kit (4-week supply) of cost-free quit smoking medication (nicotine replacement therapy, bupropion, or varenicline) and a pre-printed prescription to be filled by the patient at the end of the 4-weeks.
  Interventions: Other: cost free pharmacotherapy
- Usual Care Group (Active Comparator): Participants assigned to the prescription only usual care group received a prescription for smoking cessation pharmacotherapy to be filled at their own cost at their local community pharmacy.
  Interventions: Other: usual care

INTERVENTIONS:
Other: cost free pharmacotherapy — Participants assigned to the CF group received a starter kit (4-week supply) of cost-free quit smoking medication (nicotine replacement therapy, bupropion, or varenicline) and a pre-printed prescription to be filled by the patient at the end of the 4-weeks.
  Arms: Cost Free Pharmacotherapy
Other: usual care — Participants assigned to the prescription only usual care group received a prescription for smoking cessation pharmacotherapy to be filled at their own cost at their local community pharmacy.
  Arms: Usual Care Group

SUMMARY:
This pilot study examined the effect of providing a 4 weeks of cost free quit smoking medications to smokers identified in a stroke prevention clinic who were interested in quitting smoking compared to providing a prescription for the medication only.

DETAILED DESCRIPTION:
DESIGN: Randomized controlled trial. METHODS: All patients seen at the Ottawa Hospital Stroke Prevention Clinic were screened for smoking status, advised to quit smoking and treated using a standardized protocol including counselling and pharmacotherapy. Eligible smokers were randomly assigned to either a prescription only usual care group, or, the experimental group who received a 4-week supply of cost-free quit smoking medications and prescription for medication renewal. All patients received follow-up counselling 7-days prior to and 5, 14, 30, 60, 90, 180 days following their quit attempt. Levels of eligibility, consent, adherence and retention were used as indicators of study feasibility. The primary outcome was bio-chemically validated quit rates at 26-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible to participate in the study if they reported smoking an average of 5 or more cigarettes per day in past 3 months; were 18 years of age or older; were willing to set a quit date in the next 30 days; and were willing to use a quit smoking medication.

Exclusion Criteria:

* Patients who were unable to read and understand English or French or who had contraindications to all approved smoking cessation medications (nicotine replacement therapy, bupropion, and varenicline) were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
smoking abstinence | 6-months
  The dependent variables of primary interest were measured at 26 weeks and included: (1) bio-chemically confirmed 7-day point prevalence abstinence; and (2) continuous abstinence since TQD. Participants who were not available for follow-up were considered smokers. At the 26 week follow-up, all patients who reported being abstinent from smoking had their smoking status confirmed by measurement of a CO sample. If any CO was >10 ppm, the subject was considered a smoker.

SECONDARY OUTCOMES:
quit attempts | 6-months
  At the 26 week follow-up assessments patient quit attempts in the previous six months of 24 hours or longer were documented.
adherence with intervention | 6-months
  During the 26-week telephone follow-up assessment patient adherence with pharmacotherapy was assessed by evaluating the number of doses of pharmacotherapy consumed within the prescribed study interval. The telephone counsellor recorded the completion of all seven counselling sessions in order to assess patient adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Reid, Ph.D., Principal Investigator — Associate Director and Professor
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada